CLINICAL TRIAL: NCT06955637
Title: Comparison Between Removable Devices in Overjet Reduction: a Randomised Open Label Clinical Trial
Brief Title: Removable Devices in Overjet Reduction
Acronym: RemoDevOJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Eleonora Ortu, Researcher, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB L'Aquila 02/2021
Record Dates: First submitted 2025-04-16; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-03

CONDITIONS: Skeletal Class II Malocclusion; Dental Overjet
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elastodontic removable device (Experimental): Patients in this group will be treat with an elastodontic device adapted to the patient according to the shape of the dental arches. This device is similar to a mouthguard and embraces both dental arches. This appliance is worn overnight and the patient will be checked every month. The degree of will be taken at T0( before the start of the therapy), at T1 (after six months)and at T2 (after one month). All the dental recors will be taken by the same operator with an intraoral scanner 3D.
  Interventions: Device: dental movement
- Clear Aligners (Experimental): Patients in this group will be treat with clear aligners of the dental arches. This removable device Is transparent and covers all tooth surfaces perfectly. This appliance is 22 hours at day and the patient will be checked every month. The degree of will be taken at T0( before the start of the therapy), at T1 (after six months)and at T2 (after one month). All the dental records will be taken by the same operator with an intraoral scanner 3D.
  Interventions: Device: dental movement

INTERVENTIONS:
Device: dental movement — Possibility to reduce the protrusion of upper incisors

SUMMARY:
The goal of this clinical trial si to compare two removable devices used to treat the mandibular retrusion in growing patients.

The main questions it aims to answer are:

* the efficacy of the two devices in the reduction of the overjet
* the neuromuscolar effects developed on the stomatognatic system Participants will be instructed in the use and maintenance of the devices and will be checked every 15-30 days for one year.

ELIGIBILITY:
Inclusion Criteria:

* skeletal class II relationship,
* complete eruption of upper first premolars
* presence of unilateral or bilateral cross bite (falling within grade 3 IOTN index).

Exclusion Criteria:

* IOTN (INDEX OF ORTHODONTIC TREATMENT NEED) index > 4;
* presence of epilepsy,
* systemic disease,
* TMD, or periodontal disease;
* lack of written informed consent from a parent or legal guardian.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in the horizontal distance between the upper and lower incisors | 12 months
  To evaluate the possible reduction of the horizontal distance between the incisors of the two dental arches at two specific times

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento MESVA, L’Aquila, Italia, Italy

IPD SHARING:
Plan to Share IPD: No